CLINICAL TRIAL: NCT05205590
Title: The Impact of Coronavirus Disease 2019 (COVID-19) Pandemic on Migraine Disorder, Tension Headache and Epilepsy
Brief Title: COVID-19 Pandemic and Migraine Disorder, Tension Headache and Epilepsy
Status: Completed | Type: Observational
Sponsor: Aswan University (Other)
Responsible Party: Principal Investigator, Bastawy Al Fawal, Associate Professor, Aswan University
Other Study IDs: IRB: 547/7/21
Record Dates: First submitted 2022-01-24; First posted 2022-01-25 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non — Non

SUMMARY:
Coronavirus disease 2019 (COVID-19) caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) has already rapidly spread around the world as a pandemic after its first report in Wuhan, China on December 12th 2019 ( Holshue ML et al .,2019 ). As of December 27th 2020, there were more than 79.2 million confirmed cases and more than 1.7 million deaths caused by COVID-19 worldwide (WHO,2020).

Migraine& tension headacheare considered one of the most disabling chronic neurological diseases, and patients with migraine or tension headache are particularly vulnerable to drastic negative impacts of the pandemic. From heightened levels of psychosocial stress, social isolation , disruption of sleep and dietary habits ,to several COVID-19-specific concerns.

Normally, people with epilepsy (PWE)patients are very sensitive to different factors such as physical or emotional disturbances or environmental and lifestyle changes.Many factors can increase the risk of seizures,i.e., illness and fever, stressful events, sleep deprivation,changes in antiepileptic drugs (AED),use of proconvulsive treatments,to name a few.Some are unavoidable during a sociosanitary crisis like that currently being experienced.

Because of the rapid increase of infections, Government enacted a national state of emergency, limiting public mobility and compelling home confinement and social isolation. This national lockdown, in addition to the direct effects of COVID-19, have dramatically altered the lifestyle and normal routines of the entire population.Therefore, in addition to the risk of neurological involvement that COVID-19 itself has, during the pandemic,different circumstances may negatively impact on seizure control in PWE.

DETAILED DESCRIPTION:
Aim of the study:

This study aims to:

1. Explore the possible changes in migraine& tension headache frequency, severity during quarantine period.
2. Have a better understanding of the influence of the COVID-19 pandemic in people with epilepsy (PWE) and to assess whether there have been changes in seizure control during the current COVID-19 outbreak, exploring the possible causes of that.
3. Study lifestyle changes, emotions.
4. Assess quality of life before and after pandemic.

Inclusion criteria :

1. Patient with migraine (with and without Aura) diagnosed according to the international classification of headache disorders 3rd edition ( ICHD-3)
2. Patient with Chronic tension-type headache diagnosed according to ( ICHD-3)
3. Patient with epilepsy diagnosed according to The International League Against Epilepsy (ILAE).
4. Patients, whether they are infected or not infected with COVID-19.

Exclusion criteria :

1. Age below 20years.
2. Acute infarction or hemorrhage.
3. Inability to respond to questionnaires.
4. Severe medical illness.
5. Drug or alcohol abuse.
6. Patient with history of cerebrovascular stroke or TIA ,DM ,addiction, drugs as calcium blockers or beta blockers.

Patient & Method :

This study will be conducted at Aswan University Hospital on patients who will come to the Neuropsychiatry Clinic.

1. Patients will be asked to answer questionnaires related to their diseases e.g. change in frequency and severity during the lockdown period , compliance to treatment ,difficulty in getting medications, sleep and eating habits disturbance, work and overall worries during pandemic.
2. Depression & anxiety will be assessed before and after pandemic COVID-19 by Hamilton Anxiety and Hamilton Depression scale.(Arabic version).
3. Quality of life Questionnaire for epilepsy before and after COVID-19 pandemic.
4. Quality of life Questionnaire for Migraine before and after COVID-19 pandemic.
5. Quality of life Questionnaire for Tension headache before and after COVID-19 pandemic.

Study type : it's cross section study.

Sample type calculation:

It was carried out using G*Power 3 software . A calculated minimum sample of 300 patients will be needed to detect an effect size of 0.1 in the mean of Hamilton Depression and Anxiety Scales , with an error probability of 0.05 and 90% power on a two-tailed test.

Statistical analysis:

Data will be processed by the researchers and analyzed using IBM-SPSS 21.0 (IBM- SPSS Inc., Chicago, IL, USA) .

Descriptive statistics: means, standard deviations, and percentages will be calculated ,Test of significances: Chi-Square/Fisher's Exact tests will be used to compare the difference in distribution of frequencies among different groups.Independent t-test analysis will be carried out compare the means of dichotomous data.A significant p-value wasconsidered when it is equal or less than 0.05.

Ethical considerations:

1. Risk -benefit assessment:There is no risk on the patients included in thestudy
2. Confidentiality (dealing with data and data dissemination should be confidential):The confidentiality of patient's information willbe maintained throughout the study
3. The research procedure will be described in detailsto each patient providing the aims and outcomes of the study as described above.The acceptance to participate will be solely voluntary.
4. Informed consent:An informed consent will be obtained from all the patients,the study will be approved by ethical committee in faculty of medicine Aswan University

ELIGIBILITY:
Inclusion Criteria:

1. Patient with migraine (with and without Aura) diagnosed according to the international classification of headache disorders 3rd edition ( ICHD-3)
2. Patient with Chronic tension-type headache diagnosed according to ( ICHD-3)
3. Patient with epilepsy diagnosed according to The International League Against Epilepsy (ILAE).
4. Patients, whether they are infected or not infected with COVID-19.

Exclusion Criteria:

1. Age below 20years.
2. Acute infarction or hemorrhage.
3. Inability to respond to questionnaires.
4. Severe medical illness.
5. Drug or alcohol abuse.
6. Patient with history of cerebrovascular stroke or TIA ,DM ,addiction, drugs as calcium blockers or beta blockers.

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients presented to the Neuro-psychiatry outpatient Clinic, Aswan University Hospital
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Migraine, Tension Headache and Epilepsy due to COVID-19 pandemic | 8 months
  Frequency

CONTACTS AND LOCATIONS:
Overall Officials: Bastawy M AlFawal, MD, Principal Investigator — Aswan University
Locations (1):
- Aswan University, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Undecided